CLINICAL TRIAL: NCT05482893
Title: A Phase 1/2, Open-Label, Dose Escalation and Expansion Study With PT886 (Spevatamig) Followed by a Multi-cohorT Study in Patients With Advanced GastrIc, Gastroesophageal JuNction, Pancreatic Ductal or Biliary Tract AdEnocarcinomas of PT886, in Combination With ChemotherApy, and/or an Immune ChecKpoint Inhibitor. The TWINPEAK Study
Brief Title: Spevatamig (PT886) as Monotherapy or in Combination With Chemo and/or ICI, for the Treatment of Patients With Advanced Gastric, Gastroesophageal Junction, Pancreatic Ductal or Biliary Tract Carcinomas (the TWINPEAK Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phanes Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PT886X1101; KEYNOTE-F58 (MK-3475-F58) (Other: Merck Sharp & Dohme, LLC)
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-06

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Biliary Tract Cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel; pembrolizumab; Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): An accelerated titration design will be employed for early dose levels, followed by the standard 3+3 design at higher dose levels.
  Interventions: Drug: Spevatamig (PT886)
- Dose Expansion (Experimental): Two dose levels will be explored; the recommended dose for expansion (RDE) from Part A, and another dose level.
  Interventions: Drug: Spevatamig (PT886)
- Combination Expansion with Chemotherapy (Experimental): Part C, Cohort C1: 2L m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with Paclitaxel.
  Part C, Cohort C2: 1L m/a PDAC patients will receive Spevatamig (PT886) in combination with Gemcitabine plus nab-Paclitaxel (Abraxane).
  Part C, Cohort C3: 1L m/a PDAC patients will receive Spevatamig (PT886) in combination with Gemcitabine plus FOLFIRINOX/mFFX.
  Part C, Cohort C4: 2L BTC patients will receive PT886 in combination with SOC chemotherapy mFOLFOX6.
  Cohort C5, 1L HER2 negative PD-L1 CPS < 1 GC/GEJC patients will receive PT886 in combination with SOC chemotherapy mFOLFOX6 or CAPOX.
  Interventions: Drug: Spevatamig (PT886); Drug: Paclitaxel; Drug: Gemcitabine; Drug: Abraxane; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Capecitabine; Drug: FOLFIRINOX
- Combination Expansion with KEYTRUDA® (pembrolizumab) (Experimental): Part D, Cohort D2: Patients with m/a GC/GEJ-C, that have progressed under 1L SOC chemotherapy, and zolbetuximab, will receive Spevatamig (PT886) in combination with KEYTRUDA® (pembrolizumab).
  Part D, Cohort D3: 2L or 3L m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with KEYTRUDA® (pembrolizumab).
  Part D, Cohort D4: 1L HER2 negative m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with SOC chemotherapy and KEYTRUDA® (pembrolizumab).
  Interventions: Drug: Spevatamig (PT886); Drug: KEYTRUDA® (pembrolizumab); Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Capecitabine

INTERVENTIONS:
Drug: Spevatamig (PT886) — Spevatamig (PT886) monotherapy, a novel bispecific antibody that targets Claudin 18.2 and CD47.
Drug: Paclitaxel — Chemotherapy as a combination partner to Spevatamig (PT886) in Part C: Cohort C1
  Arms: Combination Expansion with Chemotherapy
Drug: Gemcitabine — Chemotherapy as a combination partner to Abraxane and Spevatamig (PT886) in Part C: Cohort C2
  Arms: Combination Expansion with Chemotherapy
Drug: Abraxane — Chemotherapy as a combination partner to Gemcitabine and Spevatamig (PT886) in Part C: Cohort C2
  Arms: Combination Expansion with Chemotherapy
Drug: KEYTRUDA® (pembrolizumab) — Immune checkpoint inhibitor as a combination partner to Spevatamig (PT886) in Part D: Cohort D2, D3 and D4.
  Arms: Combination Expansion with KEYTRUDA® (pembrolizumab)
Drug: Oxaliplatin — Chemotherapy as a combination partner to KEYTRUDA® (pembrolizumab) and Spevatamig (PT886) in Part D: Cohort D4
  Arms: Combination Expansion with Chemotherapy; Combination Expansion with KEYTRUDA® (pembrolizumab)
Drug: Leucovorin — Chemotherapy as a combination partner to KEYTRUDA® (pembrolizumab) and Spevatamig (PT886) in Part D: Cohort D4
  Arms: Combination Expansion with Chemotherapy; Combination Expansion with KEYTRUDA® (pembrolizumab)
Drug: Fluorouracil — Chemotherapy as a combination partner to KEYTRUDA® (pembrolizumab) and Spevatamig (PT886) in Part D: Cohort D4
  Arms: Combination Expansion with Chemotherapy; Combination Expansion with KEYTRUDA® (pembrolizumab)
Drug: Capecitabine — Chemotherapy as a combination partner to KEYTRUDA® (pembrolizumab) and Spevatamig (PT886) in Part D: Cohort D4
  Arms: Combination Expansion with Chemotherapy; Combination Expansion with KEYTRUDA® (pembrolizumab)
Drug: FOLFIRINOX — Chemotherapy as a combination partner to Spevatamig (PT886) in Part C: Cohort C3
  Arms: Combination Expansion with Chemotherapy

SUMMARY:
This is a first-in-human, Phase 1/2, open-label, dose escalation and dose expansion and combination study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of Spevatamig (PT886). Patients with the following tumor types will be eligible for screening: unresectable or metastatic gastric adenocarcinoma, gastroesophageal junction (GEJ) adenocarcinoma, biliary tract carcinoma (BTC) and pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Key Inclusion Criteria

1. 18 years or older and able to sign informed consent and comply with the protocol.
2. Measurable disease as defined by RECIST V1.1 criteria for solid tumors.
3. 3. Part A and Part B: Histologically or cytologically confirmed unresectable advanced or metastatic solid gastric, gastroesophageal junction (GEJ), biliary tract or pancreatic carcinomas previously treated for advanced (metastatic or unresectable) disease or for which treatment is not available or not tolerated.

   Part C, Cohort C1: 2L m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with Paclitaxel. Patients who are HER2 positive are eligible.

   Part C, Cohort C2: 1L m/a PDAC patients will receive Spevatamig (PT886) in combination with Gemcitabine plus nab-Paclitaxel (Abraxane).

   Part C, Cohort C3: 1L m/a PDAC patients will receive Spevatamig (PT886) in combination with Gemcitabine plus FOLFIRINOX/mFFX.

   Cohort C4: Patients with m/a BTC who have progressed on 1L SOC chemotherapy (GemCis) ± ICI and are eligible for 2L SOC FOLFOX treatment.

   Cohort C5: Patients with m/a HER2 negative GC/GEJC and present a PD-L1 CPS score of <1%, who are treatment naïve for their m/a disease and eligible for treatment with SOC chemotherapy (mFOLFOX6 or CAPOX).

   Part D, Cohort D2: Patients with m/a GC/GEJ-C, that have progressed under 1L SOC chemotherapy, and zolbetuximab, will receive Spevatamig (PT886) in combination with KEYTRUDA® (pembrolizumab).

   Part D, Cohort D3: 2L or 3L m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with KEYTRUDA® (pembrolizumab).

   Part D, Cohort D4: 1L HER2 negative m/a GC/GEJ-C patients will receive Spevatamig (PT886) in combination with SOC chemotherapy and KEYTRUDA® (pembrolizumab).
4. Biopsies:

   Able to provide a formalin fixed, paraffin embedded (FFPE) tumor tissue sample (preferably fresh biopsy or if not possible, archival tissue) to be assessed for CLDN18.2 expression and other biomarkers.

   Parts C and D: Patients must present with ≥ 10%; ≥ 2+ CLDN18.2 positive TC in their tumor tissue.
5. ECOG performance status of 0 or 1.
6. Adequate organ function confirmed at screening and within 72 hours of initiating treatment.

Key Exclusion Criteria

Patients are excluded from the study if any of the following criteria apply:

1. Women who are pregnant or lactating.
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control.
3. Has an active autoimmune disease that has required systemic treatment in the past 2 years.
4. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to study treatment.
5. Patients with a history of (non-infectious) pneumonitis that required steroids, current pneumonitis, or have a history of interstitial lung disease. History of COVID-19 pneumonia with fibrotic changes.
6. Patients with untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed (e.g., evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain/CNS metastases).
7. Prior CLDN18.2 or CD47 targeting therapies, or SIRPα (signal regulatory protein alpha) targeting agents. For Part D, Cohort D2, prior treatment with zolbetuximab is allowed.
8. Impaired cardiac function or significant diseases.
9. Prior hemolytic anemia or Evans Syndrome in the last 3 months.
10. Active gastric perforation, pyloric obstruction, complete biliary obstruction, complete or incomplete intestinal obstruction requiring clinical intervention, or pleural effusion or peritoneal effusion requiring clinical intervention.
11. Patients who have experienced any thromboembolic event such as deep vein thrombosis (DVT) or pulmonary embolism in the past 6 months.

Additional inclusion and exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicity (DLT) of Spevatamig (PT886). | Through study completion.
To determine the maximum tolerated dose (MTD) of Spevatamig (PT886). | Through study completion.
To evaluate the safety and tolerability of Spevatamig (PT886). | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of Spevatamig (PT886). | Through study completion, an average of 2 years
To evaluate the immunogenicity (ADA) of Spevatamig (PT886). | Through study completion, an average of 2 years
Preliminary Efficacy of Spevatamig (PT886). | Through study completion.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarah Cannon Research Institute (SCRI), Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Duke Cancer Center, Durham, North Carolina
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, GI Medical Oncology Dept, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin